CLINICAL TRIAL: NCT00157664
Title: Canadian Longitudinal Thrombosis in End Stage Renal Disease Pilot Study
Brief Title: Long Study - Longitudinal Thrombosis in End Stage Renal Disease
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Catherine Clase Associate Professor of Medicine, McMaster University
Organization: McMaster University (Other)
Other Study IDs: MOP - 64452
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Last update posted 2008-06-17 (Estimated); Status verified 2008-06

CONDITIONS: End Stage Renal Disease; Thrombosis; Bleeding; Cardiovascular Disease
MeSH Terms: conditions — Kidney Failure, Chronic; Thrombosis; Hemorrhage; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum and plasma
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The primary focus of this study is to collect information through diagnostic testing, blood sample analysis and patient data collection on patients starting hemodialysis to determine risk and preventative factors of bleeding and clotting events.

DETAILED DESCRIPTION:
Hemodialysis patients have a very high rate of heart attacks, strokes and amputation. These problems are caused by a blood vessel problem called atherosclerosis (hardening of the arteries), and by clotting. Clotting is also a problem in the access, which is their lifeline for hemodialysis. We have early results which show that some risk factors for clotting in the general population are common in dialysis patients. Bleeding is another significant problem within this population. In this pilot study we will measure bleeding/clotting factors in the blood of consenting patients who are just starting dialysis. We will also do special tests to show how much calcium build up and atherosclerotic build up has happened in the arteries and whether the arteries are becoming stiff. We will then follow patients for up to four years and record any health problems that might reflect bleeding, clotting or a blood vessel problem. At the end of the study, we will compare people who have had bleeding, clotting or blood vessel problem with those who have not, and learn which of the measurements predicted problems. We will go on to study potential treatments, such as anti-clotting drugs, which might prevent or delay the occurrence of such problems. This would improve the health of dialysis patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (aged > 18 years)
* Patient on hemodialysis between 30 and 90 days

Exclusion Criteria:

* Anticipated recovery of renal function (on dialysis < 90 days)
* Critical illness at time of recruitment (patients who are critically ill [ICU] when first screened, who survive to 80 days, will be rescreened and will be able to participate at that point if no longer critically ill)
* Planned live-donor renal transplant within 6 months
* Patient cannot consent due to language barrier
* Patient cannot consent due to cognitive difficulties
* Patient cannot consent due to hearing impairment
* Patient cannot consent due to speech impairment
* Patient or decision maker declines consent
* Patient is unable to give consent and no substitute decision maker is available
* Patient on dialysis longer than 90 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult subjects initiating dialysis
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2004-07; Primary Completion 2008-05 (Estimated); Study Completion 2008-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Alistair J Ingram, MD, Principal Investigator — Associate Professor, Medicine; Catherine M Clase, MD, Principal Investigator — Associate Professor, Medicine; Mark A Crowther, MD, Principal Investigator — Associate Professor, Medicine
Locations (1):
- St. Joseph's Hospital, Hamilton, Ontario, Canada